CLINICAL TRIAL: NCT02897830
Title: Evaluation of Ixazomib, Lenalidomide, Dexamethasone Induction and Extended Consolidation Followed by Lenalidomide Maintenance in Newly Diagnosed Multiple Myeloma Patients ≤65 Years Eligible for High Dose Therapy
Brief Title: Ixazomib, Lenalidomide, Dexamethasone Induction and Extended Consolidation Plus Lenalidomide Maintenance in Multiple Myeloma
Acronym: IFM2014-03
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: negatives results
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Takeda (Industry); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14 7261 03
Record Dates: First submitted 2015-07-17; First posted 2016-09-13 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study treatment (Experimental): Ixazomib, Lenalidomide, Dexamethasone Induction and extended Consolidation followed by Lenalidomide Maintenance
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — induction therapy: comprising three 28-day cycles with Ixazomib (4 mg) on Days 1, 8 and 15 plus Lenalidomide (25 mg) on Days 1 through 21 and Dexamethasone (40 mg) on Days 1, 8, 15 and 22.
  Early consolidation : (consolidation part 1) will start 2 months (-/+ 14 days) after transplantation and will comprise 2 cycles of MLN - Rd (MLN R identical to induction therapy but low dose of Dexamethasone 20mg/d once a week).
  Late consolidation (consolidation part 2) will consist in 6 additional 28-day cycles of Ixazomib (4 mg on Days 1, 8 and 15) plus Lenalidomide (25 mg on Days 1 through 21).
  Other Names: MLN 9708
Drug: Lenalidomide — induction therapy: comprising three 28-day cycles with Ixazomib (4 mg) on Days 1, 8 and 15 plus Lenalidomide (25 mg) on Days 1 through 21 and Dexamethasone (40 mg) on Days 1, 8, 15 and 22.
  Early consolidation : (consolidation part 1) will start 2 months (-/+ 14 days) after transplantation and will comprise 2 cycles of MLN - Rd (MLN R identical to induction therapy but low dose of Dexamethasone 20mg/d once a week).
  Late consolidation (consolidation part 2) will consist in 6 additional 28-day cycles of Ixazomib (4 mg on Days 1, 8 and 15) plus Lenalidomide (25 mg on Days 1 through 21).
  Maintenance therapy will start within 28 days after the last dose of Lenalidomide in last cycle of Late Consolidation: Lenalidomide 10 mg/d taken on Days 1 through 21 for thirteen 28-day cycles
  Other Names: Revlimid
Drug: Dexamethasone — induction therapy: comprising three 28-day cycles with Ixazomib (4 mg) on Days 1, 8 and 15 plus Lenalidomide (25 mg) on Days 1 through 21 and Dexamethasone (40 mg) on Days 1, 8, 15 and 22.
  Early consolidation : (consolidation part 1) will start 2 months (-/+ 14 days) after transplantation and will comprise 2 cycles of MLN - Rd (MLN R identical to induction therapy but low dose of Dexamethasone 20mg/d once a week).

SUMMARY:
Open-label study to evaluate the safety and efficacy of Ixazomib in combination with Lenalidomide and Dexamethasone in patients with newly diagnosed multiple myeloma (MM). The patient population will consist of adult men and women up to 65 years, who have a confirmed diagnosis of MM who meet eligibility criteria.

DETAILED DESCRIPTION:
Patients will receive induction therapy, comprising three cycles with Ixazomib, plus Lenalidomide and Dexamethasone.

Peripheral Blood Stem Cells (PBSC) will be mobilized within 2 weeks (+/- 1 week) after the last dose of Lenalidomide, with Cyclophosphamide plus G-CSF or Granulocyte-CSF(Colony Stimulating Factor).

Intensification: High Dose Melphalan (HDM) will be performed within 3 weeks +/- 1 week following stem cell harvest.

After Peripheral Blood Stem Cell Transplantation, patient will enter in the consolidation phase:

Early consolidation (consolidation part 1) will start 2 months after transplantation and will comprise 2 cycles of MLN - Rd (MLN R identical to induction therapy but low dose of Dexamethasone).

Late consolidation (consolidation part 2) will consist in 6 additional cycles of Ixazomib plus Lenalidomide. No Dexamethasone.

Maintenance therapy will start within 28 days after the last dose of Lenalidomide in last cycle of Late Consolidation for thirteen 28-day cycles (approximately 12 months duration) Patients will be seen at regular treatment cycle intervals while they are participating in the study.

Response will be assessed according to the International Myeloma Working Group (IMWG) criteria until disease progression. All patients will be followed for survival after progression.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma based on the new IMWG Diagnostic Criteria for plasma cells disorders
* Symptomatic myeloma with CRAB criteria
* Measurable disease requiring systemic therapy defined by serum M-component ≥ 5g/l or urine M-component ≥ 200 mg/24h or serum FLC ≥ 100 mg/l.
* Subjects must not have been treated previously with any systemic therapy for multiple myeloma.
* Eligibility for high dose therapy.
* Life expectancy ≥ 3 months
* ECOG performance status 0, 1 or 2
* Patients must meet the following clinical laboratory criteria:

  * Adequate hepatic function,
  * Absolute neutrophil count (ANC) ≥ 1.0 × 109/L within 14 days prior to enrollment.
  * Hemoglobin ≥ 8 g/dL (80 g/L) within 14 days prior to enrollment
  * Platelet count ≥ 75 × 109/L eRenal eGFR ≥ 50 mL/minute within 7 days

Exclusion Criteria:

* Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening
* Evidence of mucosal or internal bleeding and/or platelet refractory.
* Prior myeloma systemic therapy
* Major surgery within 14 days before first dose of study drug.
* Radiotherapy within 14 days before first dose of study drug.
* Corticosteroids if exceed the equivalent of 160 mg of dexamethasone within 14 days before first dose of study drug
* Central nervous system involvement
* Growth factors within 7 days of screening
* Transfusion within 7 days of screening
* Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to first dose of study drug
* Infection .
* Evidence of current uncontrolled cardiovascular conditions,
* Systemic treatment, within 14 days before first dose of study drug, with strong inhibitors of CYP1A2 , strong inhibitors of CYP3A or use of Ginkgo biloba or St. John's wort.
* Ongoing or active systemic infection, known human immunodeficiency virus (HIV) positive, known active hepatitis B virus hepatitis, or known active hepatitis C virus hepatitis and history of hepatitis B or C virus hepatitis.

  15. Co-morbid systemic illnesses or other severe concurrent disease that, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Psychiatric illness/social situation that would limit compliance with study requirements.
* Known allergy to any of the study medications,
* Contraindication to any of the required concomitant drugs
* Diagnosed or treated for another malignancy within 5 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease.
* Patient has significant neuropathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
rate of stringent complete response | 13 months
  after consolidation and before maintenance therapy

SECONDARY OUTCOMES:
Adverse events | up 60 Months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
response rates | 3 months, 5 months, 7 months, 13 months, 25 months
  response rates according to the IMWG criteria after induction, high dose Melphalan, early consolidation, late consolidation and maintenance therapy
Progression free survival | 60 months
overall survival | 60 months
Percentage of patients for whom more than 5X106 CD34 cells will be collected. | 3 months
  At stem cell harvest
Correlation between presence of deletion 17p and response rate | 60 months
  biological prognostic factors assessed at D1 influencing outcome and response rates assessed at 60th month
Correlation between presence of translocation4-14 and response rate | 60 months
  biological prognostic factors assessed at D1 influencing outcome and response rates assessed at 60th month

CONTACTS AND LOCATIONS:
Overall Officials: Michel ATTAL, MD, Principal Investigator — University Hospital, Toulouse; Murielle ROUSSEL, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hosptial Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No